CLINICAL TRIAL: NCT04844619
Title: Evaluation of Effectiveness of KDR2-2 Suspension Eyedrop on Neovascular Regression in the Treatment of Neovascular Glaucoma: an Exploratory Clinical Trial
Brief Title: KDR2-2 Suspension Eyedrop in the Treatment of Neovascular Glaucoma (KDR-NVG) Trial
Acronym: KDR-NVG
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiulan Zhang, Professor of Ophthalmology, Director of Clinical Research Center, Director of CFDA-certified Pharmaceutical Research Unit, State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021KYPJ080
Record Dates: First submitted 2021-04-13; First posted 2021-04-14 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Neovascular Glaucoma; Neovascularization
Keywords: Neovascular Glaucoma; Neovascularization; anti-VEGF; vascular endothelial growth factor
MeSH Terms: conditions — Glaucoma, Neovascular; Neovascularization, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KDR2-2 group (Experimental): The patients with NVG will receive 4.0 mg/ml or 16.0mg/ml KDR2-2 suspension eyedrop and the anti-neovascular effect of KDR2-2 would be evaluated during the follow-up visits.
  Interventions: Drug: 4mg/ml KDR2-2 suspension eyedrop; Drug: 16mg/ml KDR2-2 suspension eyedrop

INTERVENTIONS:
Drug: 4mg/ml KDR2-2 suspension eyedrop — KDR2-2 is a synthetic anti-angiogenic chemical compound with highly effective inhibition on vascular endothelial growth factor receptor-2 (VEGFR2), and an additional, moderate inhibitory effect on platelet-derived growth factor receptor β (PDGFRβ).
  KDR2-2 suspension eyedrop is developed for the treatment of iris neovascularization.
  Other Names: Low-dose KDR2-2
Drug: 16mg/ml KDR2-2 suspension eyedrop — KDR2-2 is a synthetic anti-angiogenic chemical compound with highly effective inhibition on vascular endothelial growth factor receptor-2 (VEGFR2), and an additional, moderate inhibitory effect on platelet-derived growth factor receptor β (PDGFRβ).
  KDR2-2 suspension eyedrop is developed for the treatment of iris neovascularization.
  Other Names: High-dose KDR2-2

SUMMARY:
The clinical trial is aimed to evaluate the anti-neovascular effect of KDR2-2 suspension eyedrop in the treatment of neovascular glaucoma. Fourty subjects would receive either 0.96 or 3.84 mg/per day/eye, in a QID fashion, ×7 days (those without complications can continue to 28 days). The anti-neovascular effect of KDR2-2 on iris neovascularization would be evaluated at day 1, day 7, day 14, day 28 after KDR2-2 usage.

DETAILED DESCRIPTION:
Neovascular glaucoma (NVG) has a high blinding rate and poor prognosis. Anti-glaucoma surgery is the main stake of saving visual function and relieving pain, but the proliferation of iris neovascularization (NVI) makes it difficult to treat NVG. Normally, the patients need an intravitreal injection of anti-vascular endothelial growth factor (anti-VEGF) agents prior to glaucoma surgery to control the NVI proliferation.

KDR2-2, a novel small-molecule tyrosine kinase inhibitor targeting VEGF receptor 2 (VEGFR2), has demonstrated anti-neovascular effect without obvious side-effects or complications in animal studies and a Phase I clinical trial (NCT04620109). In this study, 40 patients with NVG will be included to evaluate the effectiveness of KDR2-2 suspension eyedrop on NVI in NVG eyes. The included subjects would receive either 0.96 or 3.84 mg/day/eye, in a QID fashion, ×7 days (those without complications can continue to 28 days).

This study aims to and propose a novel, non-invasive and more compliant method for the treatment of NVG.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75;
* The best-corrected visual acuity (BCVA) of the included eyes was <0.01 (Snellen chart);
* The BCVA of the contralateral eye of the included subjects was >0.1;
* Patients with clinically diagnosed neovascular glaucoma; The diagnostic criteria for neovascularization glaucoma were as follows: Intraocular pressure > 21mmHg measured by Goldmann applanation tonometer; Neovascularization is seen in the iris or anterior chamber angle, with or without corneal edema;
* Compliance with follow up for more than 28 days and written informed consent obtained;

Exclusion Criteria:

* Intravitreal injection of anti-VEGF drugs within 3 month before enrollment;
* Participation in other clinical trials within 1 month;
* Suffering from other ocular diseases that affect ocular examinations (e.g. keratopathy, uveitis, intraocular infection, etc.);
* Those who plan to receive ocular surgery during the follow-up period;
* Premenopausal women without birth control;
* Having other systemic diseases such as severe liver and kidney function damage, cardiovascular disorders, respiratory disorders, etc.) that may affect the anti-neovascular effect of KDR2-2 or more likely to develop adverse events ;
* Systemic infections under treatment;
* Any study in which the physician believes that the patient's condition will interfere with the clinical trial (e.g., the patient is prone to stress, mood disorders, depression, etc.);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of iris neovascularization | Day 0 and 7
  Changes of the iris neovascularization using anterior photography or anterior optical coherence tomography angiography.

SECONDARY OUTCOMES:
Intraocular pressure | Day 0，7 and 28
  Measurement of intraocular pressure using non-contact tonometer or iCare tonometer
Best-corrected visual acuity | Day 0，7 and 28
  Measurement of best-corrected visual acuity with Snellen LogMAR Chart
Adverse events | Day 0，7 and 28
  Adverse events related with the anti-angiogenic effect of KDR2-2
Changes of iris neovascularization | Day 0，7 and 28
  Changes of the iris neovascularization using anterior photography or anterior optical coherence tomography angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Xiulan Zhang, MD, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No